CLINICAL TRIAL: NCT06049563
Title: Evaluation of Imaging Acquisition Protocol for the Upper Abdomen Scan on a Low Field MRI Scanner (0.4T) and Comparison of the Image Quality Obtained With Respect to the Conventional Examination Performed on a High Field MRI Scanner (1.5T)
Brief Title: Evaluation of Upper Abdomen Imaging With Low Field MRI Scanner (0.4T)
Status: Completed | Type: Observational
Sponsor: Esaote S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP000001
Record Dates: First submitted 2023-09-05; First posted 2023-09-22 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Enrolled subjects: An additional MRI scan of the upper abdomen will be performed on all the subjects with the low-field 0.4 T MRI system.
  Interventions: Diagnostic Test: Diagnostic MRI

INTERVENTIONS:
Diagnostic Test: Diagnostic MRI — MRI scan of the upper abdomen performed with the low-field 0.4T MRI system.

SUMMARY:
The goal of this observational, cross-sectional, prospective study is to compare the quality of the image obtained on the upper abdomen organs with a low-field 0.4 T MRI system with the one obtained with a high-field 1.5 T MRI system, taken as a comparator and reference device.

The study is conducted on 40 consecutive adults, not vulnerable, patients who are already scheduled for diagnostic imaging examinations on the upper abdominal organs with the reference device.

DETAILED DESCRIPTION:
The Primary endpoint of the study is to :

a) compare the image quality of the upper abdominal organs obtained with 0.4 T systems and with 1.5 T systems; This will be assessed via a noninferiority study on image quality. The image quality will be assessed by two experienced radiologists (more than 5 years' experience) and a trainee radiologist (at least 2 years) via blinded independent readings of the diagnostic images acquired both on the low-field 0.4T MRI device and on reference device e.g. the high-end 1.5T MRI device

Secondary endpoints of this study are:

1. evaluate the accuracy of representation and measurement (diameters, volumes) of the gallbladder and bile and pancreatic ducts;
2. compare the exam comfort with 0.4 T systems and with 1.5 T systems by means of questionnaires on the exam comfort provided to the subjects

ELIGIBILITY:
Inclusion Criteria:

* all subjects (in-patients or out-patients) who go to the diagnostic clinical center with the indication of performing an upper abdomen MRI examination with MRI 1.5T
* age :18 years old or higher
* the subject must be capable and willing to fulfill all study requirements

Exclusion Criteria:

* pregnancy,
* poor cooperation
* claustrophobia (only for 1.5T MRI)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in-patients or out-patients, who go to the diagnostic clinical center with the indication of performing an upper abdomen MRI examination with MRI 1.5T
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Image quality assessment | On average within 7 days from intervention
  Assess the image quality obtained with Low field 0.4 T MRI scan of the upper abdomen with the hig-field 1.5 T MRI scans of the same body part

SECONDARY OUTCOMES:
Measurements accuracy: Linear measurements | On average within 7 days from the intervention
  accuracy of the measurement: diameters of gallbladder, bile and pancreatic ducts in millimeters (mm)
Measurements accuracy: volumetric measurement | On average within 7 days from the intervention
  accuracy of the measurement: diameters of gallbladder, bile and pancreatic ducts will be combined to report the related volume in milliliters (cm^3)
Comfort of the Exam | immediately after the intervention
  Data related to the comfort of the exam are collected utilizing a survey provided to the subjects entitled "Evaluation of exam comfort". The survey reports scores on a scale. For each question the subject will assign a score ranging from 1 to 5 is assigned where value 1 represents the value corresponding to the highest level of satisfaction and the value 5 to the lowest.

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Palumbo, MD, Principal Investigator — U.O.C Radiologia II Universitaria, S. Salvatore Hospital, L'Aquila, Italy
Locations (1):
- U.O.C Radiologia II Universitaria, S. Salvatore Hospital,, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: No
There's no plan to make individual partecipant data (IPD) available to other researches

REFERENCES:
- [Background] Wacker F, Branding G, Zimmer T, Faiss S, Wolf KJ. [MR cholangiopancreatography using an open low field system of 0.2 tesla: early clinical results compared with a high field system (1.5 tesla) and ERCP]. Rofo. 1997 Dec;167(6):579-84. doi: 10.1055/s-2007-1015586. German. PMID 9465952